CLINICAL TRIAL: NCT01253044
Title: Initial Randomized Controlled Trial of Acceptance and Commitment Therapy (ACT) for Distress and Impairment in OEF/OIF Veterans
Brief Title: Acceptance and Commitment Therapy (ACT) for OEF/OIF Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Responsible Party: Principal Investigator, Ariel Lang, PhD, Professor, Veterans Medical Research Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W81XWH-08-2-0159
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Results first posted 2015-10-19 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-09

CONDITIONS: Distress; Anxiety; Depression; Postconcussive Symptoms
Keywords: OEF/OIF; Veterans; Psychotherapy
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acceptance and Commitment Therapy (Experimental): 12 weeks of individually delivered Acceptance and Commitment Therapy
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Present Centered Therapy (Active Comparator): 12 weeks of individually delivered Present Centered Therapy
  Interventions: Behavioral: Present Centered Therapy

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Acceptance and Commitment Therapy, delivered twelve 60-minute one-on-one treatment sessions over 6-10 weeks (additional weeks are permissible if needed).
  Other Names: ACT
  Arms: Acceptance and Commitment Therapy
Behavioral: Present Centered Therapy — Present Centered Therapy, delivered twelve 60-minute one-on-one treatment sessions over 6-10 weeks (additional weeks are permissible if needed).
  Other Names: PCT
  Arms: Present Centered Therapy

SUMMARY:
This trial compares two psychotherapies, Acceptance and Commitment Therapy (ACT) and Present Centered Therapy (PCT), for veterans of the conflicts in Iraq and Afghanistan. We hypothesize that ACT will be more effective than PCT at reducing emotional distress and improving functioning. We further hypothesize that both interventions will be highly acceptable to participants.

DETAILED DESCRIPTION:
The proposed study is a randomized controlled trial (RCT) of Acceptance and Commitment Therapy (ACT) as compared to a control psychotherapy, Present Centered Therapy (PCT), for individuals with distress and impairment who deployed as part of Operation Enduring Freedom and/or Operation Iraqi Freedom (OEF/OIF). ACT was selected for study because it has a number of advantages for this population. It is not tied to any particular symptom constellation, so it can be applied to a variety of presenting concerns (Hayes, Luoma, et al., 2006; Öst, 2008, Powers et al., 2009), resulting in reduced training burden for clinicians and less need for applying sequential treatments to address co-morbidities. ACT has good face validity (i.e., "it makes sense") and conveys a compelling message to young Service Members and Veterans. ACT asks individuals to move forward in accordance with one's values regardless of limitations rather than struggling against those limitations. ACT appears to be acceptable to patients (mean attrition of 15.4% in 13 RCTs (Öst, 2008). ACT is being widely disseminated without adequate evidence of its effectiveness for this important population.

ELIGIBILITY:
Inclusion Criteria:

* Previous deployment to OEF or OIF
* Current distress and impairment [at least one Diagnostic and Statistical Manual version IV (DSM-IV) anxiety or depressive disorder as determined by the Mini International Neuropsychiatric Interview (MINI) or post-concussive symptoms (PCS) as determined by a positive traumatic brain injury (TBI) screen with a score of 25 or greater on the Rivermead with distress or impairment related to PCS].
* Capable of giving informed consent.

Exclusion Criteria:

* Cognitive impairment that would interfere with treatment. Potential participants will be excluded if they screen positive for more than mild cognitive impairment on the Montreal Cognitive Assessment (MoCA; excluded if score < 26).
* Severe psychopathology (psychosis, bipolar illness, urgent suicidality or self-injurious behavior) or untreated substance dependence in the past month.
* Anticipated change in pharmacologic intervention. Patients may stay on their current medications during the study but will be asked to refrain from beginning or altering medication use during the study to the extent possible.
* Other psychotherapy focusing on the same target symptoms. Patients may attend self-help groups or treatment for other types of problems (e.g., couples counseling) but not other treatment for the same presenting problems.
* Anticipated deployment or other circumstance that would interfere with completion of all study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2010-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariel J Lang, PhD, Principal Investigator — University California San Diego
Locations (6):
- United States (6):
  - VA San Diego Healthcare System, La Jolla, California
  - Walter Reed National Military Medical Center, Washington D.C., District of Columbia
  - Togus VA Medical Center, Augusta, Maine
  - Durham VA Medical Center, Durham, North Carolina
  - Cincinnati VA Medical Center, Cincinnati, Ohio
  - VA Puget Sound Health System, Seattle, Washington

REFERENCES:
- [Derived] Bomyea J, Lang AJ, Schnurr PP. TBI and Treatment Response in a Randomized Trial of Acceptance and Commitment Therapy. J Head Trauma Rehabil. 2017 Sep/Oct;32(5):E35-E43. doi: 10.1097/HTR.0000000000000278. PMID 28060206

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acceptance and Commitment Therapy | Present Centered Therapy
Started | 80 | 80
Completed | 42 | 51
Not Completed | 38 | 29
Not completed — Lost to Follow-up | 38 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acceptance and Commitment Therapy | Present Centered Therapy | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (7.9) | 34.0 (8.1) | 34.2 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 32
  Male | 65 | 63 | 128
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 12 | 21
  Not Hispanic or Latino | 70 | 65 | 135
  Unknown or Not Reported | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 10 | 18
  White | 60 | 60 | 120
  More than one race | 8 | 5 | 13
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Brief Symptom Inventory 18 (BSI-18)
Description: To determine if receiving ACT, as compared to PCT, is associated with reduced distress as measured by the BSI-18 General Symptom Index (GSI) at the end of treatment. The BSI-18 GSI summarizes a respondent's overall level of distress. The score used in a normatively based T-score (range 1-100) calculated from the sum of responses. Higher scores are indicative of greater distress.
Time Frame: Baseline and week 12
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Acceptance and Commitment Therapy | Present Centered Therapy
Number analyzed (Participants) | 80 | 80
T-score
  Baseline | 73.3 (8.3) | 74.0 (7.7)
  Post-treatment | 65.0 (13.1) | 66.8 (10.4)
Statistical Analysis 1: Comparison: Acceptance and Commitment Therapy vs Present Centered Therapy; Test type: Superiority or Other; p = .912, MMRM

2. Secondary Outcome: Sheehan Disability Inventory
Description: To determine if receiving ACT, as compared to PCT, is associated with reduced functional impairment at the end of treatment. The score used is an average (range 0-10) of completed items, with higher scores indicating greater disability.
Time Frame: Baseline and week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acceptance and Commitment Therapy | Present Centered Therapy
Number analyzed (Participants) | 80 | 80
units on a scale
  Baseline | 6.7 (2.0) | 6.4 (1.9)
  Post-treatment | 4.9 (2.4) | 5.3 (2.2)
Statistical Analysis 1: Comparison: Acceptance and Commitment Therapy vs Present Centered Therapy; Test type: Superiority or Other; p = .273, MMRM

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Acceptance and Commitment Therapy | Present Centered Therapy
Serious Adverse Events (participants affected / at risk) | 1/80 | 3/80
Other Adverse Events (participants affected / at risk) | 0/80 | 0/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acceptance and Commitment Therapy (N=80) | Present Centered Therapy (N=80)
Nephrectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Alcohol poisoning (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidality (Psychiatric disorders) | 0 (0) | 1 (1)
Agitated altercation (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No